CLINICAL TRIAL: NCT03772561
Title: An Investigator Sponsored Phase I Study of the Safety, Tolerability and Pharmacodynamics of Escalating Doses of Combination Treatment of AZD5363 + Olaparib + Durvalumab (MEDI4736) in Patients With Advanced or Metastatic Solid Tumor Malignancies.
Brief Title: Phase I Study of AZD5363 + Olaparib + Durvalumab in Patients With Advanced or Metastatic Solid Tumor Malignancies
Acronym: MEDIPAC
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC01/01/18; 2018/00137 (Other: NHG Domain Specific Research Board)
Record Dates: First submitted 2018-12-10; First posted 2018-12-11 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Solid Tumor, Adult
Keywords: AZD5363; Olaparib; Durvalumab; Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- AZD5363+Olaparib+Durvalumab (Experimental): A traditional 3+3 design will be used during the dose escalation part of the study.
  Patients will receive AZD5363 orally twice a day 4 days-on/ 3 days-off starting 14 days prior to cycle 1 day 1 (C1D1). Olaparib continuously twice a day at 300mg and Durvalumab intravenously at 1500mg once every 4 weeks will commence at C1D1. Treatment will continue until disease progression or the development of unacceptable toxicities.
  Interventions: Drug: AZD5363+Olaparib+Durvalumab

INTERVENTIONS:
Drug: AZD5363+Olaparib+Durvalumab — Patients will receive AZD5363 orally twice a day 4 days-on/ 3 days-off starting 14 days prior to cycle 1 day 1 (C1D1). Olaparib continuously twice a day at 300mg and Durvalumab intravenously at 1500mg once every 4 weeks will commence at C1D1. Treatment will continue until disease progression or the development of unacceptable toxicities.

SUMMARY:
This is a Phase 1 dose-escalation study to evaluate the safety and tolerability of combination treatment of AZD5363 + Olaparib + Durvalumab and to determine the RP2D in patients with advanced or metastatic solid tumor malignancies.

The purpose of this trial is to determine if combination treatment of drugs, Olaparib, AZD5363 and Durvalumab has beneficial effects in advanced or metastatic cancers and to determine the effects it has on patients and their cancer.

Primary Objectives

• To evaluate the safety and tolerability of combination treatment AZD5363 + Olaparib + Durvalumab and determine the Maximum Tolerated Dose (MTD), Dose-Limiting Toxicities (DLTs), and Recommended Phase 2 Dose (RP2D) for patients with advanced or metastatic solid tumor malignancies.

Secondary Objectives

* To determine the pharmacodynamics (PDn) of combination treatment AZD5363 + Olaparib + Durvalumab in patients with advanced or metastatic solid tumor malignancies
* To describe anti-tumor response using immune RECIST of combination treatment AZD5363 + Olaparib + Durvalumab in patients with advanced or metastatic solid tumor malignancies

Exploratory Objectives

* To evaluate anti-tumour response using RECIST v1.1 for combination treatment AZD5363 + Olaparib + Durvalumab in patients with advanced or metastatic solid tumor malignancies
* To explore molecular correlates of the relationship between mutations in Akt/ PIK3CA/PTEN pathway and response to AZD5363 +Olaparib+ Durvalumab
* To understand the role of tumour microenvironment in regulation of intratumoral immune regulators (i.e. T-regulatory cells) in improving response to Durvalumab
* To understand the role of AZD5363 as an immunomodulator
* To evaluate the role of PD-1 and PDL-1 immunohistochemical and tumour MMR status in predicting response to immune check point inhibitors.

DETAILED DESCRIPTION:
This study is divided into 3 different periods: Screening, Treatment, and End of Treatment Before taking the treatment, patients will have some tests and procedures done to make sure they are eligible for the study (Screening). Then they will enter the Treatment period, where Durvalumab, Olaparib and AZD5363 will be administered to them. If they stop taking your study medication for any reason, an End of Treatment visit will be conducted within 30 days after the last doze of study medication.

Screening Assessment:

* Written Informed Consent
* Inclusion/Exclusion Criteria
* Complete Medical History
* Prior therapies and PFS on last anti-cancer therapy
* Complete Physical Examination amp; ECOG
* Standard Clinical Neurologic Examination
* BSA
* Weight
* Blood Pressure, Pulse and Temperature
* Oxygen Saturation (Pulse Oximetry)
* 12-lead Electrocardiogram
* HbA1c and fasting glucose
* Serum Chemistry (renal panel 2) amp; Serum Troponin Level
* Amylase and lipase
* Liver function test
* Serum Pregnancy Test (for women of childbearing potential)
* Thyroid function test including TSH and free T4
* Coagulation Parameters
* Chest X-ray (if clinically indicated)
* CBC with Differential
* CT or MRI Scan Tumor Measurement
* PET-CT/PET-MRI Scan Tumor Measurement (optional)
* Transthoracic Echo/ MUGA
* Baseline Symptoms
* Concomitant Medication Assessments
* Tumor Biopsy
* Fasting lipids
* Assessment for hepatitis B surface antigen, hepatitis C antibodies and HIV antibodies
* Urinalysis

Run-in Period (Day -14 until Day 0)

* Complete or Symptom Directed Physical Examination amp; ECOG
* Standard Clinical Neurologic Examination
* BSA
* Weight
* Blood Pressure, Pulse and Temperature
* 12-lead Electrocardiogram
* Serum Chemistry (renal panel 2)
* Serum Troponin Level
* Coagulation Parameters
* Liver panel including amylase and lipase
* CBC with Differential
* Oxygen Saturation (Pulse Oximetry)
* Drug Administration only for AZD5363
* Pharmacodynamics (PDn) blood
* AE Assessments
* Concomitant Medication Assessments

Cycle 1 (every week)

* Complete or Symptom Directed Physical Examination amp; ECOG
* Standard Clinical Neurologic Examination
* BSA
* Weight
* Blood Pressure, Pulse and Temperature
* HbA1c ( To be performed on cycle 1 day 1and every 12 week thereafter)
* 12-lead Electrocardiogram
* Serum Chemistry (renal panel 2)
* Serum Troponin Level
* Coagulation Parameters
* Liver panel including amylase and lipase
* CBC with Differential
* Thyroid Stimulating Hormone (TSH), ACTH (only every 4 weeks, D1 of every cycle)
* Oxygen Saturation (Pulse Oximetry)
* Drug Administration
* Pharmacodynamics (PDn)
* AE Assessments
* Concomitant Medication Assessments
* Urinalysis

Cycle 2 and Cycle 3 (every 2 weeks)

* Complete or Symptom Directed Physical Examination amp; ECOG
* Standard Clinical Neurologic Examination
* BSA
* Weight
* Blood Pressure, Pulse and Temperature
* 12-lead Electrocardiogram
* Serum Chemistry (renal panel 2)
* Liver panel including amylase and lipase
* Serum Troponin Level
* Coagulation Parameters
* CBC with Differential
* Oxygen Saturation (Pulse Oximetry)
* Drug Administration
* Pharmacodynamics (PDn) blood (Cycle 2 Day 1)
* AE Assessments
* *CT or MRI Scan Tumor Measurement (end of Cycle 2every 8 weeks in the last week of the cycle)
* Concomitant Medication Assessments
* Fasting lipids
* Urinalysis
* Transthoracic Echo/ MUGA (only if indicated)

Cycle 4 and Beyond (every 4 weeks)

* Complete or Symptom Directed Physical Examination amp; ECOG
* Weight
* Blood Pressure, Pulse and Temperature
* Standard Clinical Neurologic Examination
* Oxygen Saturation (Pulse Oximetry)
* 12-lead Electrocardiogram
* Transthoracic Echo/ MUGA (only at C4D1)
* Fasting lipids
* Serum Chemistry (renal panel 2)
* Serum Troponin Level
* Thyroid Stimulating Hormone (TSH), ACTH
* Coagulation Parameters
* CBC with Differential
* *CT or MRI Scan Tumor Measurement (end of Cycle 4 and every 8 weeks thereafter)
* Drug Administration
* *PET-CT/PET-MRI Scan Tumor Measurement (optional) (every 8 weeks)
* AE Assessments
* Concomitant Medication Assessments
* Transthoracic Echo/ MUGA (only if indicated)

Final Visit

* Complete Physical Examination amp; ECOG
* Weight
* Blood Pressure, Pulse and Temperature
* Standard Clinical Neurologic Examination
* Oxygen Saturation (Pulse Oximetry)
* 12-lead Electrocardiogram and troponin level
* Transthoracic Echo/ MUGA
* Fasting lipids
* Serum Chemistry
* Coagulation Parameters
* CBC with Differential
* Thyroid Stimulating Hormone (TSH)
* AE assessments
* Concomitant Medication Assessment

ELIGIBILITY:
Inclusion Criteria:

1. All patients must sign an informed consent in accordance with local institutional guidelines.
2. Age >= 21
3. Histologically confirmed advanced or metastatic solid tumors who have radiological evidence of progressive disease on study entry and at least 2 measurable lesions, that is deemed unlikely to benefit from further conventional therapy, or for which no standard therapy is available. Although optional, where practicable and safe, all effort should be made by the investigator to obtain serial tumour biopsies from patients enrolled.
4. Provision of an archived tumour tissue block (or at least 10 newly cut unstained slides) where such samples exist in a quantity sufficient to allow for analysis
5. Any number of prior chemotherapy regimens will be allowed and may include biologics
6. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 1;
7. Patients must have adequate bone marrow function and organ function within 2 weeks of study treatment;

   * Adequate hematologic function defined as:

     (i) platelets >= 100 x 109/L in dose escalation phase, (ii) hemoglobin >= 6.21 mmol/L or 10 g/dL, (iii) ANC >= 1.5 x 109/L, (iv) WBC >= 3.0 x 109/L. Up to 5% deviation is tolerated. Transfusions and growth factors are allowed prior to and throughout the study.
   * Hepatic function: bilirubin < 1.5 times the upper limit of normal (ULN), ALT and AST < 2.5 times ULN. For patients with hepatic metastasis ALT and AST < 5 times ULN is permitted. Up to 10% deviation is acceptable.
   * Adequate renal function: estimated creatinine clearance of >= 60 mL/min, calculated using the formula of Cockcroft and Gault: (140-Age) • Mass (kg)/(72 • creatinine mg/dL); multiply by 0.85 if female.
   * Amylase and lipase <= 1.5 x ULN;
   * Alkaline phosphatase limit <= 2.5 x ULN (<= 5 x ULN for patients with liver involvement of their cancer);
   * International normalization ratio (INR) (if not on anticoagulation therapy) and partial thromboplastin time (PTT) <= 1.5 x ULN;
   * Normal TSH and ACTH
8. Females of childbearing potential who are sexually active with a non sterilized male partner must use at least 2 highly effective method of contraception from the time of screening and must agree to continue using such precautions for 180 days after the last dose of durvalumab + any drug combination therapy or 90 days after the last dose of durvalumab monotherapy. Non-sterilized male partners of a female patient must use male condom plus spermicide throughout this period. Cessation of birth control after this point should be discussed with a responsible physician. Not engaging in sexual activity for the total duration of the drug treatment and the drug washout period is an acceptable practice; however, periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control. Female subjects should also refrain from breastfeeding throughout this period. Acceptable methods of contraception are as below:

   * Established use of oral, injected or implanted hormonal methods of contraception.
   * Placement of an intrauterine device or intrauterine system.
   * Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository.
   * Male partner sterilisation (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate).
   * True abstinence
   * It is not known whether AZD5363 has the capacity to affect the metabolism of hormonal contraceptives, so hormonal contraception should also be combined with a barrier method of contraception or patients must have evidence of non-child-bearing potential by fulfilling one of the following criteria at screening:

     * Post-menopausal: defined as aged more than 50 years and amenorrhoeic for at least 12 months following cessation of all exogenous hormonal treatments.
     * Documentation of irreversible surgical sterilisation by hysterectomy, bilateral oophorectomy or bilateral salpingectomy, but not tubal ligation
9. Non-sterilized males who are sexually active with a female partner of childbearing potential must use a male condom plus spermicide from screening through 180 days after receipt of the final dose of durvalumab + any drug combination therapy or 90 days after receipt of the final dose of durvalumab monotherapy. Not engaging in sexual activity is an acceptable practice; however, occasional abstinence, the rhythm method, and the withdrawal method are not acceptable methods of contraception. Male patients are required to use barrier methods of contraception and refrain from sperm donation throughout the study and for 180 days after the last dose of study drug. Male patients wishing to father children should be advised to arrange for freezing of sperm samples prior to the start of study treatment. Breastfeeding women are also excluded from study entry.
10. At time of registration, if the patient has had previous treatment it must have been at least 4 weeks since major surgery or radiation therapy; four weeks from any other previous anti-cancer therapy including biologics. Patients must have recovered from their treatment-related events to <=G1 with the exception of alopecia and neuropathy (<= G2 sufficient).
11. Life expectancy greater than 12 weeks
12. Patients must weigh at least 30kg
13. Patients previously treated on check point inhibitor or PARP inhibitor monotherapy will be allowed on study

Exclusion Criteria:

1. Patients with significant medical illness that in the investigator's opinion cannot be adequately controlled with appropriate therapy or would compromise the patient's ability to tolerate this therapy;
2. Radiation (except planned or ongoing palliative radiation to bone outside of the region of measurable disease) <= 3 weeks prior to starting first dose of study medication
3. Participation in another clinical study with an investigational product (IP) within 30 days of the first dose of AZD5363 or matching placebo.Treatment with any of the following:

   * Nitrosourea or mitomycin C within 6 weeks of the first dose of study treatment
   * Any investigational agents or study drugs from a previous clinical study within 30 days of the first dose of study treatment (<= 4 weeks for previous PD-1/PD-L1)
   * Any other chemotherapy, immunotherapy or anticancer agents within 3 weeks of the first dose of study treatment, except hormonal therapy with LHRH analogues for medical castration in patients with prostate cancer, which are permitted
   * Potent inhibitors or inducers or substrates of CYP3A4 or substrates of CYP2D6 within 2 weeks before the first dose of study treatment (3 weeks for St John's Wort )
4. Uncontrolled hypertension or controlled hypertension (<140/90) on more than 3 antihypertensive agents
5. Clinically significant abnormalities of glucose metabolism as defined by any of the following:

   o Diabetes mellitus type I

   o Fasting plasma glucose [fasting is defined as no calorific intake for at least 8 hours]: (i) >= 7.0mmol/L (126 mg/dL) for those patients without a pre-existing diagnosis of Type 2 diabetes mellitus (ii) >= 9.3 mmol/L (167mg/dL) for those patients with a pre-existing diagnosis of Type 2 diabetes mellitus (iii) Glycosylated haemoglobin (HbA1C) >=8.0% (63.9 mmol/mol). (iv) Requirement for insulin or more than two oral hypoglycaemic medications for routine diabetic management and control
6. Major surgical procedure within the last 28 days
7. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [eg, colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

   * Subjects with vitiligo or alopecia
   * Subjects with hypothyroidism (eg, following Hashimoto syndrome) stable on hormone replacement
   * Any chronic skin condition that does not require systemic therapy
   * Subjects without active disease in the last 5 years may be included but only after consultation with the study physician
   * Subjects with celiac disease controlled by diet alone
8. Any of the following cardiac criteria:

   * Mean resting corrected QT interval (QTc) >470 msec obtained from 3 consecutive ECGs.
   * Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG eg, complete left bundle branch block, third degree heart block
   * Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalaemia, potential for torsades de pointes, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age or any concomitant medication known to prolong the QT interval.
   * Experience of any of the following procedures or conditions in the preceding 6 months: coronary artery bypass graft, angioplasty, vascular stent, myocardial infarction, angina pectoris, congestive heart failure NYHA Grade >=2.
   * Uncontrolled hypotension - SBP <90 mmHg and/or DBP <50 mmHg.
   * Cardiac ejection fraction outside institutional range of normal or <50% (whichever is higher) as measured by echocardiogram (or MUGA scan if an echocardiogram cannot be performed or is inconclusive).Left ventricular ejection fraction (LVEF) below lower limit of normal for site.
9. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, known immunodeficiency syndrome, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease (history of interstitial lung disease will also be excluded), serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent
10. Proteinuria 3+ on dipstick analysis or >500 mg/24 hours
11. Sodium or potassium levels > CTCAE v4.1 grade 1
12. Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab. The following are exceptions to this criterion:

    * Intranasal, inhaled, topical steroids, or local steroid injections (eg, intra articular injection)
    * Systemic corticosteroids at physiologic doses not to exceed <<10 mg/day>> of prednisone or its equivalent
    * Steroids as premedication for hypersensitivity reactions (eg, CT scan premedication)
13. Female subjects who are pregnant or breastfeeding or male or female subjects of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab monotherapy.
14. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
15. History of allogeneic organ transplant
16. Known history of previous clinical diagnosis of tuberculosis
17. Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA
18. Renal failure requiring haemodialysis or peritoneal dialysis;
19. Clinically unstable, active infection requiring systemic antibiotics;
20. Concurrent cancer (except non-melanoma skin cancer or carcinoma in-situ of the cervix), unless in complete remission and off all therapy for that disease for a minimum of 3 years;
21. Patients with significantly diseased or obstructed gastrointestinal tract, malabsorption, uncontrolled vomiting or diarrhea or inability to swallow oral medications.
22. Patients with serious psychiatric or medical conditions that could interfere with treatment.
23. Patients with prior MDS/ AML
24. Require therapeutic doses of anti-coagulation with warfarin or warfarin derivatives. However, treatment with low molecular weight heparin (LMWH) is allowed.
25. Brain metastases or spinal cord compression unless asymptomatic, treated and stable off steroids and anti-convulsants for at least 1 month prior to entry into the study
26. Concurrent therapy with approved or investigational anticancer therapeutics;
27. Receipt of live attenuated vaccination within 30 days prior to study entry

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-12-03 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 5 years
  Percentage of patients who have a confirmed visit response of CR or PR.
Best objective response | 5 years
  Calculated as the best response recorded from date the combination treatment started for each patient.

CONTACTS AND LOCATIONS:
Overall Officials: David SP Tan, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ibrahim YH, Garcia-Garcia C, Serra V, He L, Torres-Lockhart K, Prat A, Anton P, Cozar P, Guzman M, Grueso J, Rodriguez O, Calvo MT, Aura C, Diez O, Rubio IT, Perez J, Rodon J, Cortes J, Ellisen LW, Scaltriti M, Baselga J. PI3K inhibition impairs BRCA1/2 expression and sensitizes BRCA-proficient triple-negative breast cancer to PARP inhibition. Cancer Discov. 2012 Nov;2(11):1036-47. doi: 10.1158/2159-8290.CD-11-0348. Epub 2012 Aug 22. PMID 22915752
- [Background] Yap TA, Sandhu SK, Carden CP, de Bono JS. Poly(ADP-ribose) polymerase (PARP) inhibitors: Exploiting a synthetic lethal strategy in the clinic. CA Cancer J Clin. 2011 Jan-Feb;61(1):31-49. doi: 10.3322/caac.20095. Epub 2011 Jan 4. PMID 21205831